CLINICAL TRIAL: NCT06244472
Title: Towards a New Generation of Magnetoencephalographs: Evaluation of the FYNA Research (Mag4Health 48 Sensors MEG's Name) System (Full-head Magnetoencephalographs System With Optically Pumped Magnetometers)
Brief Title: A New Generation of Magnetoencephalographs for High Speed Functional Brain Imaging
Acronym: DEMAGUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL23_0425; 2023-A01173-42 (Other: ID-RCB)
Record Dates: First submitted 2024-01-05; First posted 2024-02-06 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Mild Concussion; Healthy Volunteers
Keywords: Magnetoencephalographs optically pumped magnetometers (MEG OPM); Brain activity; Neuroimaging
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: In healthy subjects, we will test our hypotheses in three independent experiments (20 subjects per experiment), covering an important part of the current field of use of MEG in auditory, visual, motor and somaesthetic modalities. Subjects will have the opportunity to participate in one, two or all three experiments, as they wish.
  In adults with mild traumatic brain injury, we will test our hypotheses using resting-state recording (20 subjects).
  For all the tasks, we will carry out an acquisition with the 275-sensor SQUID (Superconducting Quantum Interference Devices) MEG system from the MEG department at CERMEP (Centre d'Etude et de Recherche Multimodal Et Pluridisciplinaire) in Lyon, and a similar acquisition with the FYNA Research system.
  If the subject has no anatomical MRI (Magnetic resonance imaging), a 3D anatomical MRI (15-minute acquisition time) on a 1.5 Tesla MRI will be performed after the last MEG examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy subjects (Experimental): Healthy volunteers aged between 18 and 70 years, without neurological or psychiatric or sleep disorders
  Interventions: Device: Experiment 1: visual and auditory attention task; Device: Experiment 2: language production and rest tasks; Device: Experiment 3: visuo-motor task
- Subjects with concussion (Experimental): Male athletes volunteers with concussion aged between 18 and 40 years, without neurological or psychiatric or sleep disorders other than cerebral concussion.
  Interventions: Device: Experiment 4: brain activity at rest

INTERVENTIONS:
Device: Experiment 1: visual and auditory attention task — We will use the FYNA Research system on 20 healthy volunteers with a visual and auditory attention task to evaluate the system's performance in recording brain signals complex frequency content.
  Arms: Healthy subjects
Device: Experiment 2: language production and rest tasks — We will use the FYNA Research system on 20 healthy healthy volunteers with a language production task to assess the system's functional mapping capabilities and a resting task to assess the system's ability to identify resting networks.
  Arms: Healthy subjects
Device: Experiment 3: visuo-motor task — We will use the FYNA Research system in 20 healthy volunteers with a visuo-motor task to evaluate the system's performance in recording brain signals when the subject moves, inducing perturbations that affect the classical system (loss of spatial precision) and the FYNA Research system (low-frequency artifacts).
  Arms: Healthy subjects
Device: Experiment 4: brain activity at rest — We will be using the FYNA Research system on 20 concussed male athletes volunteers to assess the system's ability to detect modulations in the frequency content of resting brain activity.
  Arms: Subjects with concussion

SUMMARY:
The goal is to perform a first evaluation of the capabilities of a new generation of non-invasive magnetoencephalography whole head device using optically pumped magnetometers using Helium 4 as the sensitive element (OPM He4) to record brain magnetic activities. The investigators will record 1) healthy subjects stimulated with visual, auditory, somesthesic and motor stimuli and 2) athletes who suffered a mild concussion. The main hypothesis is that the OPM magnetoencephalographs (MEG) system will be able to detect brain activity. The secondary hypothesis is that the data recorded with the OPM MEG system will allow to reconstruct maps of the brain activity. To test the main hypothesis, they will compare the signal to noise ratio of brain activities between a classical MEG system and the new OPM He4 MEG. The secondary hypothesis will be tested through a comparison of the maps of brain activity obtained thanks to the data recorded with a classical MEG system and the new OPM He4 MEG.

ELIGIBILITY:
Healthy volunteers:

Inclusion Criteria:

* Age 18 to 70
* Strongly motivated to participate to the study
* Signed informed consent for the study

Exclusion Criteria:

* major cognitive deficit and unable to understand the instructions
* previous neurology or psychiatric or sleep pathologies
* Woman with a positive pregnancy test during the inclusion.
* Subjects under guardianship, curatorship or safeguard of justice protection
* Subjects deprived of their liberty
* Subject not affiliated to a social security system.
* Subject with common contraindications to MEG and MRI examination :

  * Metal in the body incompatible with performance of the examination (pacemaker, implantable pump, neurostimulator, cochlear implant, auditory prothesis, metalic prothesis, intracerebral clip, implantable defibrillator, any metalic parts in the brain or upper part of the body, ventriculoperitoneal valve, dental appliance or steel pivot for root canal, ferromagnetic foreign body in the upper part of the upper part of the body)
  * Claustrophobia

Subjects who suffered a mild concussion:

Inclusion Criteria:

* Male aged from 18 to 40
* Strongly motivated to participate to the study
* Signed informed consent for the study
* Mild concussion confirmed by the club doctor and a neurologist neurologist in the three weeks preceding the experiment

Exclusion Criteria:

* major cognitive deficit and unability to understand the instructions
* previous neurology or psychiatric or sleep pathologies except mild concussion
* Woman with a positive pregnancy test during the inclusion.
* Subjects under guardianship, curatorship or safeguard of justice protection
* Subjects deprived of their liberty
* Subject not affiliated to a social security system
* Subject with common contraindications to MEG and MRI examination :

  * Metal in the body incompatible with performance of the examination (pacemaker, implantable pump, neurostimulator, cochlear implant, auditory prothesis, metalic prothesis, intracerebral clip, implantable defibrillator, any metalic parts in the brain or upper part of the body, ventriculoperitoneal valve, dental appliance or steel pivot for root canal, ferromagnetic foreign body in the upper part of the upper part of the body)
  * Claustrophobia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Signal to Noise Ratio comparison between classical MEG and FYNA Research for the visual stimulations | Visit 2 (during the intervention, scheduled from 1 to 30 days from inclusion visit V1).
  The signal to noise ratio of normal (SNR) brain activity following a visual stimulus will be computed with respect to the pre-stimulus baseline -100 milliseconds to -10 milliseconds.
  We will compare the SNRs obtained with the classical MEG system serving as a reference and the SNRs obtained with the new OPM He4 MEG through the group of healthy volunteers for this given stimulus.
Signal to Noise Ratio comparison between classical MEG and FYNA Research for the auditory stimulations | Visit 2 (during the intervention, scheduled from 1 to 30 days from inclusion visit V1).
  The signal to noise ratio of normal (SNR) brain activity following an auditory stimulus will be computed with respect to the pre-stimulus baseline -100 milliseconds to -10 milliseconds .
  We will compare the SNRs obtained with the classical MEG system serving as a reference and the SNRs obtained with the new OPM He4 MEG through the group of healthy volunteers for this given stimulus.
Signal to Noise Ratio comparison between classical MEG and FYNA Research for the somesthesia stimulations | Visit 2 (during the intervention, scheduled from 1 to 30 days from inclusion visit V1).
  The signal to noise ratio of normal (SNR) brain activity following a somesthetic stimulus will be computed with respect to the pre-stimulus baseline -100 milliseconds to -10 milliseconds .
  We will compare the SNRs obtained with the classical MEG system serving as a reference and the SNRs obtained with the new OPM He4 MEG through the group of healthy volunteers for this given stimulus.
Signal to Noise Ratio comparison between classical MEG and FYNA Research for the motor stimulations | Visit 2 (during the intervention, scheduled from 1 to 30 days from inclusion visit V1).
  The signal to noise ratio of normal (SNR) brain activity following a motor stimulus will be computed with respect to the pre-stimulus baseline -100 milliseconds to -10 milliseconds .
  We will compare the SNRs obtained with the classical MEG system serving as a reference and the SNRs obtained with the new OPM He4 MEG through the group of healthy volunteers for this given stimulus.
Signal to Noise Ratio comparison between classical MEG and FYNA Research for the rest activity | Visit 2 (during the intervention, scheduled from 1 to 30 days from inclusion visit V1).
  The signal to noise ratio of normal (SNR) brain activity at rest will be computed with respect to the pre-stimulus baseline -100 milliseconds to -10 milliseconds .
  We will compare the SNRs obtained with the classical MEG system serving as a reference and the SNRs obtained with the new OPM He4 MEG through the group of male athletes with concussion.

SECONDARY OUTCOMES:
Correlation of maps of brain activity | Visit 2 (during the intervention, scheduled from 1 to 30 days from inclusion visit V1).
  We will report the spatial correlation between the maps computed with the classical MEG system and the ones computed with the new OPM He4 MEG. The classical MEG will serve as a reference.
  Healthy volunteers solely.
Evaluation of the comfort of the subject during the optically pumped magnetometers (OPM) He4 MEG recordings through a short verbal questionnaire (scores of the absolute and relative comfort scales). | 5 minutes after the end the recording session
  The evaluation will be done verbally through a short questionnaire. This questionnaire evaluates the overall comfort of the OPM system with two questions: 1) An evaluation of the overall comfort thanks to a scale with five steps from very uncomfortable to very comfortable and 2) A comparison with the classical MEG system thanks to a 5 steps scale from much less comfortable than the classical MEG system to much more comfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Julien JUNG, MD, Principal Investigator — Service d'Epilepsie et Explorations fonctionnelles neurologiques,Hôpital Neurologique P. Wertheimer, Groupement Hospitalier Est, HCL
Locations (2):
- France (2):
  - Service de Neurologie Fonctionnelle et d'Epileptologie, Hôpital Neurologique Pierre Wertheimer, Hospices Civils de Lyon, Bron
  - Centre Orthopédique Paul Santy, Lyon

IPD SHARING:
Plan to Share IPD: No